CLINICAL TRIAL: NCT07000851
Title: Neuroinflammation, White Matter Integrity, AD Biomarkers and Pathology in Corticobasal Syndrome
Brief Title: Imaging Studies in Corticobasal Syndrome
Acronym: I-CAN
Status: Recruiting | Type: Observational
Sponsor: Jennifer Whitwell (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Jennifer Whitwell, Associate Consultant II, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 24-007544; 1R01AG087140-01A1 (NIH)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Cortico Basal Degeneration; Corticobasal Syndrome; Corticobasal Syndrome(CBS); Corticobasal Degeneration; Corticobasal Degeneration (CBD); Corticobasal Syndrome (CBS)
Keywords: neurodegeneration; neurodegenerative disease; cbs; cbd; corticobasal syndrome; corticobasal degeneration
MeSH Terms: conditions — Corticobasal Degeneration; Nerve Degeneration; Neurodegenerative Diseases; Color Vision Defects

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Corticobasal Syndrome: patients diagnosed with cbs
  Interventions: Diagnostic Test: C-11 ER176 Radiotracer; Diagnostic Test: C-11 PiB; Diagnostic Test: AV1451 Tau
- Healthy Control: Healthy Control Volunteer
  Interventions: Diagnostic Test: C-11 ER176 Radiotracer; Diagnostic Test: C-11 PiB; Diagnostic Test: AV1451 Tau

INTERVENTIONS:
Diagnostic Test: C-11 ER176 Radiotracer — PET scan looking for inflammation
Diagnostic Test: C-11 PiB — PET scan looking for amyloid protein
Diagnostic Test: AV1451 Tau — Pet scan looking for Tau protein

SUMMARY:
The primary goal of this study is to investigate inflammation and white matter damage in corticobasal syndrome and determine whether these processes are related to each other. The investigator's will address our goal by using neuroimaging and blood plasma biomarkers, as well as molecular pathology.

DETAILED DESCRIPTION:
Corticobasal syndrome (CBS) is a neurodegenerative disorder characterized by cognitive and behavioral change, as well as asymmetric parkinsonism, dystonia, myoclonus, and limb apraxia. Emerging evidence suggests neuroinflammation plays a key role in the pathogenesis of neurodegenerative disease, including the 4R tauopathies and AD, and neuroinflammation has been linked mechanistically to damage of the white matter. The primary goal of this study is to investigate inflammation and white matter damage using imaging and blood samples.

The investigator's will use the PET ligand 11C-ER176 to assess patterns of neuroinflammation in the brain and Neurite Orientation Dispersion and Density Imaging (NODDI) to measure white matter microstructure, including axonal density and alignment. The investigator's will also investigate blood plasma metrics, including neurofilament light chain and plasma glial fibrillary acidic protein (GFAP) that measure neuroaxonal injury and astrogliosis, and inflammation and tau metrics. The investigator's will employ beta-amyloid (A) and tau (T) PET to subdivide the CBS patients into those with biomarker AD (A+T+, CBS-AD) and those without biomarker AD (CBS-4R). The investigator's will also compare these groups to disease controls with typical amnestic biomarker AD (Amn-AD) and healthy controls (HC) that have previously been recruited for other grants (existing data collected under approved IRBs).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Meet possible or probable CBS criteria

Exclusion Criteria:

* Subjects will be excluded if MRI is contraindicated (due to implanted device, severe claustrophobia, etc)
* Subjects will be excluded if they have a concurrent illnesses or structural abnormality that could account for the CBS syndrome
* Subjects will be excluded if they have a mutation in the progranulin gene
* Subjects will excluded if they have received anti-Aβ therapy
* Women who are pregnant will be excluded
* Subjects will be excluded if they are actively taking daily anti-inflammatory medications (NSAIDs, corticosteriods, etc)
* Subjects will be excluded if they have generalized inflammatory condition and treatment with immunosuppressive, corticoid/glucocorticoid, steroidal or non-steroidal anti-inflammatory medication within 2 weeks of scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who meet criteria are eligible to participate
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2030-03-30 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
The investigators will use C-11 ER176 PET imaging to evaluate neuroinflammation and white matter integrity in CBS | approximately 4-5 years into study visits
  Measure whether regional patterns of ER176-PET uptake and white matter microstructure abnormalities using NODDI differ between CBS-4R, CBS-AD, Amn-AD, and HC.

SECONDARY OUTCOMES:
the investigators will use blood samples to assess inflammatory and tau blood plasma metrics in CBS. | approximately 4-5 years into study visits
  Measure whether plasma metrics differ between CBS-4R, CBS-AD, Amn-AD, and HC.

OTHER OUTCOMES:
The investigators will use MR imaging to compare regional markers of inflammation, white matter integrity and tau burden in autopsy tissue from patients with CBS from two different 4R tauopathies and CBS-AD. | Approximately 8-10 years after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Whitwell, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No